CLINICAL TRIAL: NCT00417183
Title: Randomized Controlled Trial Comparing the Long GnRH Agonist Protocol and the Flexible GnRH Antagonist Protocol of Ovarian Stimulation in Normal Responders
Brief Title: Comparison of the Long GnRH Agonist Protocol and the Flexible GnRH Antagonist Protocol of Ovarian Stimulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eugonia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: long vs flexible
Record Dates: First submitted 2006-12-22; First posted 2006-12-29 (Estimated); Last update posted 2006-12-29 (Estimated); Status verified 2006-12

CONDITIONS: Infertility
Keywords: GnRH antagonist; GnRH agonist; Long protocol; Flexible
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate; ganirelix

INTERVENTIONS:
Drug: Arvekap 0.1 mg (Triptorelin, Ipsen, France)
Drug: Ganirelix 0.25 (Orgalutran, Organon, The Netherlands)

SUMMARY:
The purpose of this study is to compare the efficacy of two controlled ovarian stimulation protocols, the GnRH agonist protocol, widely known as the "long" protocol, and the flexible GnRH antagonist protocol, in terms of pregnancy rates and embryological data, in infertile patients receiving IVF treatment.

DETAILED DESCRIPTION:
The formulation of controlled ovarian stimulation protocols is one of the primary reasons for the successful development of IVF. The "long" GnRH agonist protocol, also known as the gold standard, has been widely used with considerable success. More recently, on the other hand, GnRH antagonist provide a new promising approach for endogenous gonadotrophin suppression by blocking the GnRH receptor. There is conflicting data in the literature regarding the relative merits of the two ovarian stimulation protocols.

COMPARISON: Pregnancy rates and embryological data will by assessed in IVF patients treated with either the "long" GnRH agonist (Arvekap) or the flexible GnRH antagonist (Ganirelix) protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39 years
* Body mass index 18-29 kg/m2
* Menstrual cycle from 24-35 days
* Normal basal FSH (<10 IU/ml)
* Normal basal LH (<10 IU/ml)
* Normal basal estradiol (<80 pg/ml)

Exclusion Criteria:

* Poor responder patients
* Polycystic ovaries

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2005-09; Study Completion 2007-06

PRIMARY OUTCOMES:
Ongoing pregnancy per embryo transfer

SECONDARY OUTCOMES:
Biochemical pregnancy per embryo transfer
Clinical pregnancy per embryo transfer
Embryological data

CONTACTS AND LOCATIONS:
Overall Officials: Tryfon Lainas, PhD, Principal Investigator — Eugonia
Locations (1):
- Eugonia, Athens, Greece

REFERENCES:
- [Background] Lainas T, Zorzovilis J, Petsas G, Stavropoulou G, Cazlaris H, Daskalaki V, Lainas G, Alexopoulou E. In a flexible antagonist protocol, earlier, criteria-based initiation of GnRH antagonist is associated with increased pregnancy rates in IVF. Hum Reprod. 2005 Sep;20(9):2426-33. doi: 10.1093/humrep/dei106. Epub 2005 Jun 9. PMID 15946995